CLINICAL TRIAL: NCT03152097
Title: Targeting FMO-Mediated TMAO Formation in Kidney Disease (TMAO) Study
Acronym: TMAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Thomas Nolin, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: PRO16090410
Record Dates: First submitted 2017-05-04; First posted 2017-05-12 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Kidney Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Kidney Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): This crossover design will include 4 weeks of diindolylmethane and 4 weeks of matching placebo assignment.
  Interventions: Dietary Supplement: Commercially available Diindolylmethane; Other: Placebo
- Commercially available Diindolylmethane (Experimental): This crossover design will include 4 weeks of diindolylmethane and 4 weeks of matching placebo assignment.
  Interventions: Dietary Supplement: Commercially available Diindolylmethane; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Commercially available Diindolylmethane — Commercially available Diindolylmethane is a compound derived from cruciferous vegetables (e.g. broccoli)
Other: Placebo — A matching placebo capsule will be compounded by the UPMC Investigational Drug Service

SUMMARY:
The project will investigate the modulation of flavin-containing monooxygenase (FMO) formation of the CVD risk factor trimethylamine-N-oxide (TMAO) in patients with kidney disease.

DETAILED DESCRIPTION:
Twelve patients with stage 3 to 4 kidney disease will receive an intervention for four weeks and a matching placebo in a crossover study design. Reduction of serum TMAO from baseline to end of intervention will be the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age, but not more than 75 years of age at the time of enrollment.
2. Must be able to provide signed and dated informed consent.
3. Medical diagnosis of chronic kidney disease (eGFR ≤ 60 ml/min/1.73m2 )

Exclusion Criteria:

1. Vital signs outside of acceptable range at Screening Visit
2. Use of any of the following drugs within the last 3 months:

   Systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral); oral, intravenous, intramuscular, nasal or inhaled corticosteroids; cytokines; methotrexate or immunosuppressive cytotoxic agents; anti-diarrheal agents, bile acid sequestrants.
3. Consuming commercial probiotics including tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component. Ordinary dietary components such as fermented beverages/milks, yogurts, foods do not apply.
4. Chronic, clinically significant hepatic abnormality (i.e. elevated 3X ULN ALT/AST), as determined by medical history or physical examination.
5. History of cancer except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision.
6. Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.
7. Recent history of chronic alcohol consumption defined as more than five 1.5-ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day.
8. Any confirmed or suspected condition/state of immunosuppression or immunodeficiency.
9. History of active uncontrolled gastrointestinal disorders or diseases including: Inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis; irritable bowel syndrome (IBS) (moderate-severe); persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated); chronic constipation. Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
10. Patient who may be pregnant or lactating.
11. Not willing to abstain from cruciferous vegetable (i.e. cabbage, brussels sprouts, garden cress, mustard greens, turnips, broccoli, collard greens , cauliflower, kale) consumption.
12. Current smoking.
13. Unwilling or unable to adhere to study procedures or instructions.
14. Patients taking any of the following medications, methimazole, alosetron, duloxetine, ramelteon, tasimelteon, theophylline, tizanidine, clozapine, pirfenidone and ramosetron.
15. Allergies to corn or soy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
TMAO | 12 weeks.
  Serum TMAO concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Nolin, PharmD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No